CLINICAL TRIAL: NCT04025424
Title: Observational Study of Genetic Predictors of Efficiency and Safety of Immune Checkpoints Inhibitors in Patients With Different Malignancies (ICIPRESIST-0519)
Brief Title: Genetic Predictors of Efficiency and Safety of ICIs in Patients With Different Malignancies (ICIPRESIST-0519)
Acronym: ICIPRESIST19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Igor Samoylenko, MD, PhD, Principal Investigator, Senior Researcher, Tumor biotherpay Department, Russian Academy of Medical Sciences
Other Study IDs: ICIPRESIST-052019
Record Dates: First submitted 2019-07-17; First posted 2019-07-18 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Melanoma; Squamous Cell Lung Cancer; Uveal Melanoma; Hodgkin Lymphoma
MeSH Terms: conditions — Melanoma; Uveal Melanoma; Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Tumor blocks and blood DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Skin melanoma, retrospective: * 1) Clinically and morphologically verified diagnosis of skin melanoma or melanoma metastases without an identified primary lesion;
  * 2) The availability of basic clinical information about the patient and the course of his illness;
  Interventions: Genetic: Genetic tests of the available tumor and plasma samples
- Hodgkin disease, retrospective: * 1) Clinically and morphologically verified diagnosis of Hodgkin disease (any histological variant);
  * 2) The availability of basic clinical information about the patient and the course of his illness;
  Interventions: Genetic: Genetic tests of the available tumor and plasma samples
- Uveal melanoma, retrospective: * 1) Clinically and morphologically verified diagnosis of uveal melanoma (any histological variant);
  * 2) The availability of basic clinical information about the patient and the course of his il
  Interventions: Genetic: Genetic tests of the available tumor and plasma samples
- Skin melanoma, proscpective: * 1) Clinically and morphologically verified diagnosis of metastatic melanoma;
  * 2) The availability of basic clinical information about the patient and the course of his illness;
  Interventions: Genetic: Genetic tests of the available tumor and plasma samples
- Lung cancer, procpective: * 1) Clinically and morphologically verified diagnosis of metastatic or inoperable squamous cell lung cancer;
  * 2) The availability of basic clinical information about the patient and the course of his illness;
  * 3) The presence of indications for therapy with a PD-1 or PD-L1 inhibitor in the standard dosage in monotherapy;
  Interventions: Genetic: Genetic tests of the available tumor and plasma samples

INTERVENTIONS:
Genetic: Genetic tests of the available tumor and plasma samples — Only available samples or samples obtainted for other reasons will be used for molecular testing. No special intervention is preplanned

SUMMARY:
This is a multicenter, non-interventional, retrospective study (with two prospective cohorts), including previously treated patients with melanoma, squamous cell lung cancer in the late stages (inoperable or metastatic) and Hodgkin disease at any stages.

The duration of the follow-up will be 12-60 months. Data from medical records will be retrospectively collected at different points in time. The first data extraction will consist of collecting data from the initial level (before treatment with immune checkpoints inhibitors (anti-PD1 / PDl1) before the end of the recruitment period for this study (up to 3 years of follow-up). Two additional annual data collections are planned for display additional follow-up and data for patients who will survive.

ELIGIBILITY:
Inclusion Criteria:

To participate in this study, the patient must meet the following criteria:

* At least 2 injections (or 10 weeks) of ICI (PD1, PDl1 blockers, including but not limited to such drugs as nivolumab, pembrolizumab, prolglimab, atezolizumab, avelumab, durvalumab, spratalizumab)
* Deceased patients meet the criteria; signing the informed consent of the legal representative of the deceased patient is not required

Specific inclusion criteria for individual cohorts:

* Cohort 1 (retrospective cohort of skin melanoma patients)

  * 1) Clinically and morphologically verified diagnosis of skin melanoma or melanoma metastases without an identified primary focus;
  * 2) The availability of basic clinical information about the patient and the course of his illness;
  * 3) Therapy with a PD-1 or PD-L1 inhibitor in the standard dosage in monotherapy (at least 2 injections);
  * 4) Evaluation of the effect of immunotherapy
  * 5) Availability of tumor material (paraffin blocks) for morphological, immunohistochemical and molecular genetic studies, obtained no earlier than 24 months. before initiating therapy with a PD-1 or PD-L1 inhibitor;
  * 8) Patient-signed informed consent in case the patient is alive
* Cohort 2 (Hodjkin disease - retrospective)

  * 1) Clinically and morphologically verified diagnosis of Hodgkin disease (any histological variant);
  * 2) The availability of basic clinical information about the patient and the course of his illness;
  * 3) Availability of tumor material (paraffin blocks) for morphological, immunohistochemical and molecular genetic studies;
  * 4) Patient signed informed consent.
* Cohort 3 (Uveal melanoma - retro)

  * 1) Clinically and morphologically verified diagnosis of uveal melanoma (any histological variant);
  * 2) The availability of basic clinical information about the patient and the course of his illness;
  * 3) Availability of tumor material (paraffin blocks) for morphological, immunohistochemical and molecular genetic studies;
  * 4) Patient signed informed consent.
* Cohort 4 (melanoma of the skin - prospective)

  * 1) Clinically and morphologically verified diagnosis of metastatic melanoma;
  * 2) The availability of basic clinical information about the patient and the course of his illness;
  * 3) Indications for therapy with a PD-1 or PD-L1 inhibitor in the standard dosage in monotherapy;
  * 4) The possibility of including the patient in the present study before the first course of immunotherapy;
  * 5) Availability of tumor material (paraffin blocks and histological glass preparations) for morphological, immunohistochemical and molecular genetic studies obtained no earlier than 2 years before the planned start of immunotherapy with a standard PD-1 inhibitor;
  * 6) Separate patient consent to a repeated biopsy of the tumor focus before the planned start of immunotherapy with a PD-1 or PD-L1 inhibitor, if the existing tumor material was obtained earlier than 2 years before the planned start of immunotherapy
  * 7) Availability of samples of biological fluids collected before the start of immunotherapy and after the first course of immunotherapy for molecular genetic studies of circulating tumor DNA;
  * 8) Evaluation of the effect of therapy in the framework of local practice in accordance with the criteria of RECIST 1.1
  * 9) Signed by the patient informed consent to participate in the study.
* Cohort 5 (squamous cell lung cancer - prospective)

  * 1) Clinically and morphologically verified diagnosis of metastatic or inoperable squamous cell lung cancer;
  * 2) The availability of basic clinical information about the patient and the course of his illness;
  * 3) The presence of indications for therapy with a PD-1 or PD-L1 inhibitor in the standard dosage in monotherapy;
  * 4) The possibility of including the patient in the present study before the first course of immunotherapy;
  * 5) Availability of tumor material (paraffin blocks) for morphological, immunohistochemical and molecular genetic research, obtained no earlier than 2 years before the planned start of immunotherapy with a standard PD-1 inhibitor;
  * 6) Separate patient consent to a repeated biopsy of the tumor focus before the planned start of immunotherapy with a PD-1 or PD-L1 inhibitor, if the existing tumor material was obtained earlier than 2 years before the planned start of immunotherapy
  * 7) Availability of samples of biological fluids collected before the start of immunotherapy and after the first course of immunotherapy for molecular genetic studies of circulating tumor DNA;
  * 8) Evaluation of the effect of therapy in the framework of local practice in accordance with the criteria of RECIST 1.1
  * 9) Signed by the patient informed consent to participate in the study.

Exclusion Criteria:

* Cohort 1 (retrospective cohort of skin melanoma patients)

  - 1) It is not allowed to conduct other immunotherapy (anti-CTLA4, vaccines, etc.) to patients before the course of therapy with a PD-1 or PD-L1 inhibitor in a standard dosage in monotherapy
* Cohort 2 (Hodgkin disease - retrospective)
* no special exclusion criteria
* Cohort 3 (Uveal melanoma - retro)

  - No special exclusion criteria.
* Cohort 4 (melanoma of the skin - prospective)

  * 1) It is not allowed to include patients who have previously undergone other immunotherapy (anti-CTLA4, vaccines, etc.) before the course of therapy with the PD-1 or PD-L1 inhibitor in the standard dosage in monotherapy
  * 2) It is not allowed to include patients who are scheduled for combination immunotherapy (anti-PD1 + anti-CTLA4, vaccines, etc.) after inclusion in this study
* Cohort 5 (squamous cell lung cancer - prospective)

  * 1) It is not allowed to include patients who have previously undergone other immunotherapy (anti-CTLA4, vaccines, etc.) before the course of therapy with the PD-1 or PD-L1 inhibitor in the standard dosage in monotherapy
  * 2) It is not allowed to include patients who are scheduled for combination immunotherapy (anti-PD1 + anti-CTLA4, vaccines, etc.) after inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target sample consists of approximately 350 treated patients, treatment of patients with melanoma, squamous cell lung cancer in the late stages (inoperable or metastatic) and Hodgkin dsisease, who met the criteria.
  The current study will be conducted in selected research centers where at least 5 patients are treated with blockers of immune checkpoints during the quarter (3 months) in the period from 2015 to 2019. In each research center, patients will be identified that meet the inclusion criteria, based on the lists of patients who received therapy with blockers of immune checkpoints in specific research centers. The study is conducted only in centers located in Russia.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) of patients receiving immune checkpoint blockers (PD1 / PDl1 blockers) in the first and subsequent treatment lines in patients with metastatic or unresectable melanoma, lung cancer and lymphoma granulomatosis | dec 2021
  Overall survival (OS) will be calculated and presented in graphical form using the method of the product of Kaplan-Meier limits. The report will include a median of C with corresponding bilateral values of 95% CI. The proportion of patients who survive at certain points in time (1, 2, and 3 years), as well as the corresponding bilateral values of 95% CI, will be evaluated and reported.
incidence and severity of all adverse events (AEs) in patients receiving immune checkpoint blockers (PD1 / PDl1 blockers) in the first and subsequent treatment lines in patients with metastatic or unresectable melanoma, lung cancer and lymphoma. | dec 2021

OTHER OUTCOMES:
progression-free survival (PFS) in patients receiving immune checkpoint blockers (PD1 / PDl1 blockers) in the first and subsequent treatment lines in patients with metastatic or unresectable melanoma, lung cancer and Hodgkin disease | dec 2021
response rate in patients receiving immune checkpoint blockers (PD1 / PDl1 blockers) in the first and subsequent treatment lines in patients with metastatic or unresectable melanoma, lung cancer and Hodgkin disease | dec 2021
Development of predictive molecular testing tools | dec 2021
  The predictive power parameters of the predictive tools being developed will be generalized using descriptive statistics methods. The significance of the results of the qualitative tests will be assessed using Fisher's two-sided exact test. The optimal threshold values for quantitative tests will be evaluated using the ROC curve method, and for the mutational load, the four squares method of Abeshouse, 2017 will also be calculated. using the proportional Cox test.

CONTACTS AND LOCATIONS:
Locations (1):
- N.N. Blokhin Russian Cancer Research Center, Moscow, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided